CLINICAL TRIAL: NCT05894694
Title: Survival Benefit of Compound Kushen Injection in Treatment of Advanced Colorectal Cancer Based on Real World Registration Platform
Brief Title: Survival Benefit of Compound Kushen Injection in the Treatment of Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Jie Li, Vice President, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-063-KY
Record Dates: First submitted 2023-04-24; First posted 2023-06-08 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Advanced Colorectal Carcinoma
Keywords: Compound kushen Injection; Traditional Chinese medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- first-line scheme + compound kushen injection (Experimental): Compound Kushen injection+first-line regimen (FOLFOX/FOLFIRI/CAPEOX± Cetuximab/bevacizumab)+
  Interventions: Drug: first-line scheme+compound kushen injection
- first-line scheme (Other): first-line regimen (FOLFOX/FOLFIRI/CAPEOX± Cetuximab/bevacizumab)
  Interventions: Drug: palliative care group first-line scheme

INTERVENTIONS:
Drug: first-line scheme+compound kushen injection — FOLFOX/FOLFIRI/CAPEOX± Cetuximab/bevacizumab+compound kushen injection Compound Kushen injection: intravenous infusion, 20ml at a time, diluted with 200ml sodium chloride injection, once a day, each cycle of chemotherapy should reach the cumulative dose of 200ml.
  Arms: first-line scheme + compound kushen injection
Drug: palliative care group first-line scheme — FOLFOX/FOLFIRI/CAPEOX± Cetuximab/bevacizumab
  Arms: first-line scheme

SUMMARY:
To clarify the effectiveness and safety of compound kushen injection in the treatment of advanced colorectal cancer.

DETAILED DESCRIPTION:
This study include a multi-center, randomized, parallel controlled clinical trial. The randomized clinical trial will enroll approximately 320 patients. Participants will be randomly divided into experimental (n=160) and control groups (n=160). Patients in the experimental group was treated with first-line scheme + compound kushen injection. Patients in the control group will receive first-line scheme. The primary endpoint is PFS. The research protocol was approved by the relevant ethics committees, and the study was conducted according to the Declaration of Helsinki and Good Clinical Practice guidelines. Patients gave written informed consent to participate in the trial.

ELIGIBILITY:
Inclusion Criteria:

① Patients with advanced CRC confirmed by pathology or cytology and receiving first-line therapy;② Aged ≥ 18 years old, male or female;③ ECOG score 0-2 points;④ Expected survival ≥ 3 months;⑤ According to RECIST1.1 criteria, at least one detectable lesion;⑥ Voluntarily join the study, sign informed consent, compliance with good cooperation with follow-up.

Exclusion Criteria:

* Combined with other malignant primary tumors;

  * Immunohistochemistry/polymerase chain reaction/second-generation sequencing results suggest MSI-H/dMMR patients;

    * Patients with recurrence and metastasis within 6 months after radical tumor surgery;

      * Patients who have previously or are undergoing cancer immunotherapy ; Patients undergoing radiation therapy;

        * Pregnant or lactating women; women of childbearing age and their spouses can not take effective contraceptive measures during and within 6 months after the end of clinical study; ⑥ Psychiatric patients; ⑦ Patients with severe, uncontrolled organic disease or infection, such as decompensated heart, lung, kidney failure caused by intolerance to chemotherapy; ⑧ Patients who have received clinical trials of small molecule drugs within 28 days or received clinical trials of large molecule drugs within 3 months; ⑨ Patients who are known to be allergic to or intolerant of study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | The time from randomization to tumor progression or death in patients, whichever came first, assessed up to 24 months
  Progression Free Survival

SECONDARY OUTCOMES:
OS | The time from randomization to death from any cause after enrollment, whichever occurs first, assessed up to 24 months
  Overall survival
1-year survival rate | The proportion of patients with survival period of more than 1 year accounted for the total patients from the beginning of enrollment treatment
  The probability of patients surviving more than 1 year after treatment
1-year PFS rate | The proportion of patients with tumor progression or death from enrollment.
  the proportion of the total patients who does not with tumor progression or death within 1 year from enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Guang 'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu J, Ge Y, Zhu G, Gao R, Zhu X, Zhang Y, Li J. Combination of Compound Kushen injection with first-line treatment versus first-line treatment alone for advanced colorectal cancer: a study protocol for a multicenter, openlabel, randomized controlled trial. BMC Complement Med Ther. 2024 Dec 31;24(1):429. doi: 10.1186/s12906-024-04725-6. PMID 39741233